CLINICAL TRIAL: NCT06146595
Title: Prevalence Study of Attention Deficit Hyperactivity Disorder and Its Comorbidities Among a Sample of Primary School Students in New Valley Governorate
Brief Title: Prevalence of Attention Deficit Hyperactivity Disorder and Its Comorbidities
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmood Mohammed Yosry Abdelsatar Mohammed, assistant lecturer, Assiut University
Other Study IDs: ADHD and its comorbidity
Record Dates: First submitted 2023-11-16; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Estimate the prevalence of attention deficit hyperactivity disorder and comorbid psychiatric disorder among primary school students in New Valley governorate.

DETAILED DESCRIPTION:
ADHD (attention deficit hyperactivity disorder) is a common neurodevelopmental disorder characterized by hyperactivity, impulsivity, and inattention. Its prevalence ranges between 5.9 and 7.1% worldwide. Etiology of ADHD included combinations of genetic, neurological, and environmental factors. ADHD is more often a complex disorder with a high rate of associated comorbid conditions. Comorbid conditions are prevalent among people with ADHD and increase its burden and complexity of management. Children with ADHD are at a higher risk than children without ADHD for developing other psychiatric disorders. Most children with ADHD also have at least one comorbid condition, the presence of which contributes to poorer long-term outcomes. The pattern of comorbidities is influenced by age and sex; externalizing disorders are more common in younger ages and male participants, in contrast, internalizing disorders are more prevalent among older ages and female participants. Comorbidity involving ADHD and learning disorders is frequent, ranging from 25 to 40%. Other disorders likely to co-occur with ADHD are: bipolar disorders (11-75%), tic disorders (20%), obsessive compulsive disorders (6-15%). Children with ADHD may show several motor problems: longer and more variable reaction times, increased variability in speed and less accurate response reengagement, and impaired orienting responses, and increased number of responses with very long reaction times. Neurological soft sign have been associated with inattention and behavior difficulties for decades. Some researchers argue that these signs should be included in the diagnosis of ADHD.

ELIGIBILITY:
Inclusion Criteria:

Age: 6-17 years. Sex: both sexes will be included in the study.

Exclusion Criteria:

Age: less than 6 years or more than 17 years. Patients with major neurological deficits, cerebral palsy. Patient who refusing to participate in the study or their caregiver refusing to give informed consent. Mentally retarded children.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: primary school students in New Valley governorate
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Detect the prevalence of attention deficit hyperactivity disorder among primary school students in New Valley governorate | Baseline
  the child and his parents will be subjected to special psychiatric interview sheet designed at child psychiatric unit at Assiut university hospital for collecting detailed psychiatric history of the child and assessment of the child through a detailed interview including mental state examination and neurological examination.also the child will be subjected to Conner's Parent Rating Scale-revised (L).

SECONDARY OUTCOMES:
Detect comorbid psychiatric disorder among ADHD primary school student in New Valley governorate. | Baseline
  the child will be subjected to Child behavior checklist (CBCL), parent form

REFERENCES:
- [Result] Belanger SA, Andrews D, Gray C, Korczak D. ADHD in children and youth: Part 1-Etiology, diagnosis, and comorbidity. Paediatr Child Health. 2018 Nov;23(7):447-453. doi: 10.1093/pch/pxy109. Epub 2018 Oct 24. PMID 30681669
- [Result] Willcutt EG. The prevalence of DSM-IV attention-deficit/hyperactivity disorder: a meta-analytic review. Neurotherapeutics. 2012 Jul;9(3):490-9. doi: 10.1007/s13311-012-0135-8. PMID 22976615
- [Result] Becker SP, Langberg JM, Evans SW. Sleep problems predict comorbid externalizing behaviors and depression in young adolescents with attention-deficit/hyperactivity disorder. Eur Child Adolesc Psychiatry. 2015 Aug;24(8):897-907. doi: 10.1007/s00787-014-0636-6. Epub 2014 Oct 31. PMID 25359419
- [Result] Mohammadi MR, Zarafshan H, Khaleghi A, Ahmadi N, Hooshyari Z, Mostafavi SA, Ahmadi A, Alavi SS, Shakiba A, Salmanian M. Prevalence of ADHD and Its Comorbidities in a Population-Based Sample. J Atten Disord. 2021 Jun;25(8):1058-1067. doi: 10.1177/1087054719886372. Epub 2019 Dec 13. PMID 31833803
- [Result] Tung I, Li JJ, Meza JI, Jezior KL, Kianmahd JS, Hentschel PG, O'Neil PM, Lee SS. Patterns of Comorbidity Among Girls With ADHD: A Meta-analysis. Pediatrics. 2016 Oct;138(4):e20160430. doi: 10.1542/peds.2016-0430. Epub 2016 Sep 21. PMID 27694280
- [Result] Yoshimasu K, Barbaresi WJ, Colligan RC, Voigt RG, Killian JM, Weaver AL, Katusic SK. Childhood ADHD is strongly associated with a broad range of psychiatric disorders during adolescence: a population-based birth cohort study. J Child Psychol Psychiatry. 2012 Oct;53(10):1036-43. doi: 10.1111/j.1469-7610.2012.02567.x. Epub 2012 May 31. PMID 22647074
- [Result] Gillberg C, Gillberg IC, Rasmussen P, Kadesjo B, Soderstrom H, Rastam M, Johnson M, Rothenberger A, Niklasson L. Co-existing disorders in ADHD -- implications for diagnosis and intervention. Eur Child Adolesc Psychiatry. 2004;13 Suppl 1:I80-92. doi: 10.1007/s00787-004-1008-4. PMID 15322959
- [Result] Cardo E, Casanovas S, de la Banda G, Servera M. [Soft neurological signs: are they of any value in the assessment and diagnosis of attention deficit hyperactivity disorder?]. Rev Neurol. 2008;46 Suppl 1:S51-4. Spanish. PMID 18302123
- [Result] Johansen EB, Aase H, Meyer A, Sagvolden T. Attention-deficit/hyperactivity disorder (ADHD) behaviour explained by dysfunctioning reinforcement and extinction processes. Behav Brain Res. 2002 Mar 10;130(1-2):37-45. doi: 10.1016/s0166-4328(01)00434-x. PMID 11864716
- [Result] Spencer TJ, Biederman J, Mick E. Attention-deficit/hyperactivity disorder: diagnosis, lifespan, comorbidities, and neurobiology. J Pediatr Psychol. 2007 Jul;32(6):631-42. doi: 10.1093/jpepsy/jsm005. Epub 2007 Jun 7. PMID 17556405
- [Result] Jensen CM, Steinhausen HC. Comorbid mental disorders in children and adolescents with attention-deficit/hyperactivity disorder in a large nationwide study. Atten Defic Hyperact Disord. 2015 Mar;7(1):27-38. doi: 10.1007/s12402-014-0142-1. Epub 2014 Jun 19. PMID 24942707